CLINICAL TRIAL: NCT06046248
Title: Phase II Trial of Belumosudil and Rituximab for the Primary Treatment of Extensive Chronic Graft-versus-host Disease
Brief Title: Belumosudil and Rituximab for Primary Treatment of Chronic Graft-Versus-Host-Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1385
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Belumosudil Plus Rituximab (Experimental): Belumosudil plus Rituximab
  Interventions: Drug: Belumosudil; Drug: Rituximab

INTERVENTIONS:
Drug: Belumosudil — 200mg PO QD x 24 cycles (28-day cycle)
Drug: Rituximab — 375mg/m2 IV Q1 week x 4 weeks, then Q3 months x4 doses

SUMMARY:
This is an open-label, Phase 2 study designed to evaluate the safety and efficacy of belumosudil and rituximab as primary treatment of cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* First episode of systemic immunosuppression-requiring cGVHD, defined as classic cGVHD by the NIH consensus criteria (without features or characteristics of aGVHD)
* Previously untreated, defined by having received <10 days of corticosteroids or alternative systemic immunosuppressive agent started specifically for a new diagnosis of cGVHD
* KPS >/= 70%
* Adequate hematologic function independent of platelet transfusion and G-CSF for at least 7 days prior to study entry: ANC >750 cells/mm3; Platelets >30,000 cells/mm#

Exclusion Criteria:

* Late persistent or recurrent aGVHD
* Active uncontrolled infection
* History of HIV infection
* Active HBV or HCV infection. Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative PCR result before enrollment. Those who are PCR positive will be excluded.
* Calculated CrCl <30mL/min
* AST and/or ALT >5x ULN or direct bilirubin >3x ULN
* Cardiac ejection fraction <40% or history of uncontrolled cardiac arrhythmias
* Has received more than one allogeneic transplant prior to the occurrence of cGVHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who achieve partial and complete responses after treatment | 2 years

SECONDARY OUTCOMES:
Length of time patients remain on corticosteroid treatment | 2 years
Number of patients who had treatment-related adverse events using CTCAE v5 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Solomon, MD, Principal Investigator — BMTGA/Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abou-Mourad YR, Lau BC, Barnett MJ, Forrest DL, Hogge DE, Nantel SH, Nevill TJ, Shepherd JD, Smith CA, Song KW, Sutherland HJ, Toze CL, Lavoie JC. Long-term outcome after allo-SCT: close follow-up on a large cohort treated with myeloablative regimens. Bone Marrow Transplant. 2010 Feb;45(2):295-302. doi: 10.1038/bmt.2009.128. Epub 2009 Jul 13. PMID 19597425
- [Result] Bhatia S, Francisco L, Carter A, Sun CL, Baker KS, Gurney JG, McGlave PB, Nademanee A, O'Donnell M, Ramsay NK, Robison LL, Snyder D, Stein A, Forman SJ, Weisdorf DJ. Late mortality after allogeneic hematopoietic cell transplantation and functional status of long-term survivors: report from the Bone Marrow Transplant Survivor Study. Blood. 2007 Nov 15;110(10):3784-92. doi: 10.1182/blood-2007-03-082933. Epub 2007 Aug 1. PMID 17671231
- [Result] Schmitz N, Eapen M, Horowitz MM, Zhang MJ, Klein JP, Rizzo JD, Loberiza FR, Gratwohl A, Champlin RE; International Bone Marrow Transplant Registry; European Group for Blood and Marrow Transplantation. Long-term outcome of patients given transplants of mobilized blood or bone marrow: A report from the International Bone Marrow Transplant Registry and the European Group for Blood and Marrow Transplantation. Blood. 2006 Dec 15;108(13):4288-90. doi: 10.1182/blood-2006-05-024042. Epub 2006 Aug 31. PMID 16946302
- [Result] Higman MA, Vogelsang GB. Chronic graft versus host disease. Br J Haematol. 2004 May;125(4):435-54. doi: 10.1111/j.1365-2141.2004.04945.x. PMID 15142114
- [Result] Koc S, Leisenring W, Flowers ME, Anasetti C, Deeg HJ, Nash RA, Sanders JE, Witherspoon RP, Storb R, Appelbaum FR, Martin PJ. Therapy for chronic graft-versus-host disease: a randomized trial comparing cyclosporine plus prednisone versus prednisone alone. Blood. 2002 Jul 1;100(1):48-51. doi: 10.1182/blood.v100.1.48. PMID 12070007
- [Result] Vogelsang GB. How I treat chronic graft-versus-host disease. Blood. 2001 Mar 1;97(5):1196-201. doi: 10.1182/blood.v97.5.1196. PMID 11222360
- [Result] Ratanatharathorn V, Ayash L, Lazarus HM, Fu J, Uberti JP. Chronic graft-versus-host disease: clinical manifestation and therapy. Bone Marrow Transplant. 2001 Jul;28(2):121-9. doi: 10.1038/sj.bmt.1703111. PMID 11509929
- [Result] Sutherland HJ, Fyles GM, Adams G, Hao Y, Lipton JH, Minden MD, Meharchand JM, Atkins H, Tejpar I, Messner HA. Quality of life following bone marrow transplantation: a comparison of patient reports with population norms. Bone Marrow Transplant. 1997 Jun;19(11):1129-36. doi: 10.1038/sj.bmt.1700806. PMID 9193757
- [Result] Chiodi S, Spinelli S, Ravera G, Petti AR, Van Lint MT, Lamparelli T, Gualandi F, Occhini D, Mordini N, Berisso G, Bregante S, Frassoni F, Bacigalupo A. Quality of life in 244 recipients of allogeneic bone marrow transplantation. Br J Haematol. 2000 Sep;110(3):614-9. doi: 10.1046/j.1365-2141.2000.02053.x. PMID 10997973
- [Result] Fraser CJ, Bhatia S, Ness K, Carter A, Francisco L, Arora M, Parker P, Forman S, Weisdorf D, Gurney JG, Baker KS. Impact of chronic graft-versus-host disease on the health status of hematopoietic cell transplantation survivors: a report from the Bone Marrow Transplant Survivor Study. Blood. 2006 Oct 15;108(8):2867-73. doi: 10.1182/blood-2006-02-003954. Epub 2006 Jun 20. PMID 16788100
- [Result] Kiss TL, Abdolell M, Jamal N, Minden MD, Lipton JH, Messner HA. Long-term medical outcomes and quality-of-life assessment of patients with chronic myeloid leukemia followed at least 10 years after allogeneic bone marrow transplantation. J Clin Oncol. 2002 May 1;20(9):2334-43. doi: 10.1200/JCO.2002.06.077. PMID 11981005
- [Result] Stewart BL, Storer B, Storek J, Deeg HJ, Storb R, Hansen JA, Appelbaum FR, Carpenter PA, Sanders JE, Kiem HP, Nash RA, Petersdorf EW, Moravec C, Morton AJ, Anasetti C, Flowers ME, Martin PJ. Duration of immunosuppressive treatment for chronic graft-versus-host disease. Blood. 2004 Dec 1;104(12):3501-6. doi: 10.1182/blood-2004-01-0200. Epub 2004 Aug 3. PMID 15292060
- [Result] Duell T, van Lint MT, Ljungman P, Tichelli A, Socie G, Apperley JF, Weiss M, Cohen A, Nekolla E, Kolb HJ. Health and functional status of long-term survivors of bone marrow transplantation. EBMT Working Party on Late Effects and EULEP Study Group on Late Effects. European Group for Blood and Marrow Transplantation. Ann Intern Med. 1997 Feb 1;126(3):184-92. doi: 10.7326/0003-4819-126-3-199702010-00002. PMID 9027268
- [Result] Socie G, Stone JV, Wingard JR, Weisdorf D, Henslee-Downey PJ, Bredeson C, Cahn JY, Passweg JR, Rowlings PA, Schouten HC, Kolb HJ, Klein JP. Long-term survival and late deaths after allogeneic bone marrow transplantation. Late Effects Working Committee of the International Bone Marrow Transplant Registry. N Engl J Med. 1999 Jul 1;341(1):14-21. doi: 10.1056/NEJM199907013410103. PMID 10387937
- [Result] Sullivan KM, Witherspoon RP, Storb R, Weiden P, Flournoy N, Dahlberg S, Deeg HJ, Sanders JE, Doney KC, Appelbaum FR, et al. Prednisone and azathioprine compared with prednisone and placebo for treatment of chronic graft-v-host disease: prognostic influence of prolonged thrombocytopenia after allogeneic marrow transplantation. Blood. 1988 Aug;72(2):546-54. PMID 3042041
- [Result] Syrjala KL, Chapko MK, Vitaliano PP, Cummings C, Sullivan KM. Recovery after allogeneic marrow transplantation: prospective study of predictors of long-term physical and psychosocial functioning. Bone Marrow Transplant. 1993 Apr;11(4):319-27. PMID 8485479
- [Result] Wingard JR, Piantadosi S, Vogelsang GB, Farmer ER, Jabs DA, Levin LS, Beschorner WE, Cahill RA, Miller DF, Harrison D, et al. Predictors of death from chronic graft-versus-host disease after bone marrow transplantation. Blood. 1989 Sep;74(4):1428-35. PMID 2670000
- [Result] Champlin RE, Passweg JR, Zhang MJ, Rowlings PA, Pelz CJ, Atkinson KA, Barrett AJ, Cahn JY, Drobyski WR, Gale RP, Goldman JM, Gratwohl A, Gordon-Smith EC, Henslee-Downey PJ, Herzig RH, Klein JP, Marmont AM, O'Reilly RJ, Ringden O, Slavin S, Sobocinski KA, Speck B, Weiner RS, Horowitz MM. T-cell depletion of bone marrow transplants for leukemia from donors other than HLA-identical siblings: advantage of T-cell antibodies with narrow specificities. Blood. 2000 Jun 15;95(12):3996-4003. PMID 10845940
- [Result] Pavletic SZ, Carter SL, Kernan NA, Henslee-Downey J, Mendizabal AM, Papadopoulos E, Gingrich R, Casper J, Yanovich S, Weisdorf D; National Heart, Lung, and Blood Institute Unrelated Donor Marrow Transplantation Trial. Influence of T-cell depletion on chronic graft-versus-host disease: results of a multicenter randomized trial in unrelated marrow donor transplantation. Blood. 2005 Nov 1;106(9):3308-13. doi: 10.1182/blood-2005-04-1614. Epub 2005 Jul 26. PMID 16046530
- [Result] Miklos DB, Kim HT, Zorn E, Hochberg EP, Guo L, Mattes-Ritz A, Viatte S, Soiffer RJ, Antin JH, Ritz J. Antibody response to DBY minor histocompatibility antigen is induced after allogeneic stem cell transplantation and in healthy female donors. Blood. 2004 Jan 1;103(1):353-9. doi: 10.1182/blood-2003-03-0984. Epub 2003 Sep 25. PMID 14512314
- [Result] Miklos DB, Kim HT, Miller KH, Guo L, Zorn E, Lee SJ, Hochberg EP, Wu CJ, Alyea EP, Cutler C, Ho V, Soiffer RJ, Antin JH, Ritz J. Antibody responses to H-Y minor histocompatibility antigens correlate with chronic graft-versus-host disease and disease remission. Blood. 2005 Apr 1;105(7):2973-8. doi: 10.1182/blood-2004-09-3660. Epub 2004 Dec 21. PMID 15613541
- [Result] Canninga-van Dijk MR, van der Straaten HM, Fijnheer R, Sanders CJ, van den Tweel JG, Verdonck LF. Anti-CD20 monoclonal antibody treatment in 6 patients with therapy-refractory chronic graft-versus-host disease. Blood. 2004 Oct 15;104(8):2603-6. doi: 10.1182/blood-2004-05-1855. Epub 2004 Jul 13. PMID 15251978
- [Result] Cutler C, Miklos D, Kim HT, Treister N, Woo SB, Bienfang D, Klickstein LB, Levin J, Miller K, Reynolds C, Macdonell R, Pasek M, Lee SJ, Ho V, Soiffer R, Antin JH, Ritz J, Alyea E. Rituximab for steroid-refractory chronic graft-versus-host disease. Blood. 2006 Jul 15;108(2):756-62. doi: 10.1182/blood-2006-01-0233. Epub 2006 Mar 21. PMID 16551963
- [Result] Okamoto M, Okano A, Akamatsu S, Ashihara E, Inaba T, Takenaka H, Katoh N, Kishimoto S, Shimazaki C. Rituximab is effective for steroid-refractory sclerodermatous chronic graft-versus-host disease. Leukemia. 2006 Jan;20(1):172-3. doi: 10.1038/sj.leu.2403996. No abstract available. PMID 16239908
- [Result] Ratanatharathorn V, Ayash L, Reynolds C, Silver S, Reddy P, Becker M, Ferrara JL, Uberti JP. Treatment of chronic graft-versus-host disease with anti-CD20 chimeric monoclonal antibody. Biol Blood Marrow Transplant. 2003 Aug;9(8):505-11. doi: 10.1016/s1083-8791(03)00216-7. PMID 12931119
- [Result] Zaja F, Bacigalupo A, Patriarca F, Stanzani M, Van Lint MT, Fili C, Scime R, Milone G, Falda M, Vener C, Laszlo D, Alessandrino PE, Narni F, Sica S, Olivieri A, Sperotto A, Bosi A, Bonifazi F, Fanin R; GITMO (Gruppo Italiano Trapianto Midollo Osseo). Treatment of refractory chronic GVHD with rituximab: a GITMO study. Bone Marrow Transplant. 2007 Aug;40(3):273-7. doi: 10.1038/sj.bmt.1705725. Epub 2007 Jun 4. PMID 17549053
- [Result] Cutler C, Kim HT, Bindra B, Sarantopoulos S, Ho VT, Chen YB, Rosenblatt J, McDonough S, Watanaboonyongcharoen P, Armand P, Koreth J, Glotzbecker B, Alyea E, Blazar BR, Soiffer RJ, Ritz J, Antin JH. Rituximab prophylaxis prevents corticosteroid-requiring chronic GVHD after allogeneic peripheral blood stem cell transplantation: results of a phase 2 trial. Blood. 2013 Aug 22;122(8):1510-7. doi: 10.1182/blood-2013-04-495895. Epub 2013 Jul 16. PMID 23861248
- [Result] Sauter CS, Barker JN, Lechner L, Zheng J, Devlin SM, Papadopoulos EB, Perales MA, Jakubowski AA, Goldberg JD, Koehne G, Ceberio I, Giralt S, Zelenetz AD, Moskowitz CH, Castro-Malaspina H. A phase II study of a nonmyeloablative allogeneic stem cell transplant with peritransplant rituximab in patients with B cell lymphoid malignancies: favorably durable event-free survival in chemosensitive patients. Biol Blood Marrow Transplant. 2014 Mar;20(3):354-60. doi: 10.1016/j.bbmt.2013.11.029. Epub 2013 Dec 4. PMID 24315843
- [Result] Solomon SR, Sizemore CA, Ridgeway M, Zhang X, Smith J, Brown S, Holland HK, Morris LE, Bashey A. Corticosteroid-Free Primary Treatment of Chronic Extensive Graft-versus-Host Disease Incorporating Rituximab. Biol Blood Marrow Transplant. 2015 Sep;21(9):1576-82. doi: 10.1016/j.bbmt.2015.04.023. Epub 2015 May 16. PMID 25985915
- [Result] Solomon SR, Sizemore CA, Ridgeway M, Zhang X, Brown S, Holland HK, Morris LE, Solh M, Bashey A. Safety and efficacy of rituximab-based first line treatment of chronic GVHD. Bone Marrow Transplant. 2019 Aug;54(8):1218-1226. doi: 10.1038/s41409-018-0399-7. Epub 2018 Dec 5. PMID 30518977
- [Result] Zanin-Zhorov A, Weiss JM, Nyuydzefe MS, Chen W, Scher JU, Mo R, Depoil D, Rao N, Liu B, Wei J, Lucas S, Koslow M, Roche M, Schueller O, Weiss S, Poyurovsky MV, Tonra J, Hippen KL, Dustin ML, Blazar BR, Liu CJ, Waksal SD. Selective oral ROCK2 inhibitor down-regulates IL-21 and IL-17 secretion in human T cells via STAT3-dependent mechanism. Proc Natl Acad Sci U S A. 2014 Nov 25;111(47):16814-9. doi: 10.1073/pnas.1414189111. Epub 2014 Nov 10. PMID 25385601
- [Result] Zeiser R, Blazar BR. Pathophysiology of Chronic Graft-versus-Host Disease and Therapeutic Targets. N Engl J Med. 2017 Dec 28;377(26):2565-2579. doi: 10.1056/NEJMra1703472. No abstract available. PMID 29281578
- [Result] Flynn R, Paz K, Du J, Reichenbach DK, Taylor PA, Panoskaltsis-Mortari A, Vulic A, Luznik L, MacDonald KK, Hill GR, Nyuydzefe MS, Weiss JM, Chen W, Trzeciak A, Serody JS, Aguilar EG, Murphy WJ, Maillard I, Munn D, Koreth J, Cutler CS, Antin JH, Ritz J, Waksal SD, Zanin-Zhorov A, Blazar BR. Targeted Rho-associated kinase 2 inhibition suppresses murine and human chronic GVHD through a Stat3-dependent mechanism. Blood. 2016 Apr 28;127(17):2144-54. doi: 10.1182/blood-2015-10-678706. Epub 2016 Mar 16. PMID 26983850
- [Result] Riches DW, Backos DS, Redente EF. ROCK and Rho: Promising therapeutic targets to ameliorate pulmonary fibrosis. Am J Pathol. 2015 Apr;185(4):909-12. doi: 10.1016/j.ajpath.2015.01.005. Epub 2015 Feb 14. PMID 25687558
- [Result] Knipe RS, Tager AM, Liao JK. The Rho kinases: critical mediators of multiple profibrotic processes and rational targets for new therapies for pulmonary fibrosis. Pharmacol Rev. 2015;67(1):103-17. doi: 10.1124/pr.114.009381. PMID 25395505
- [Result] Cutler C, Lee SJ, Arai S, Rotta M, Zoghi B, Lazaryan A, Ramakrishnan A, DeFilipp Z, Salhotra A, Chai-Ho W, Mehta R, Wang T, Arora M, Pusic I, Saad A, Shah NN, Abhyankar S, Bachier C, Galvin J, Im A, Langston A, Liesveld J, Juckett M, Logan A, Schachter L, Alavi A, Howard D, Waksal HW, Ryan J, Eiznhamer D, Aggarwal SK, Ieyoub J, Schueller O, Green L, Yang Z, Krenz H, Jagasia M, Blazar BR, Pavletic S. Belumosudil for chronic graft-versus-host disease after 2 or more prior lines of therapy: the ROCKstar Study. Blood. 2021 Dec 2;138(22):2278-2289. doi: 10.1182/blood.2021012021. Erratum In: Blood. 2022 Mar 17;139(11):1772. doi: 10.1182/blood.2022015598. PMID 34265047
- [Result] Weinstein JS, Hernandez SG, Craft J. T cells that promote B-Cell maturation in systemic autoimmunity. Immunol Rev. 2012 May;247(1):160-71. doi: 10.1111/j.1600-065X.2012.01122.x. PMID 22500839
- [Result] Flynn R, Du J, Veenstra RG, Reichenbach DK, Panoskaltsis-Mortari A, Taylor PA, Freeman GJ, Serody JS, Murphy WJ, Munn DH, Sarantopoulos S, Luznik L, Maillard I, Koreth J, Cutler C, Soiffer RJ, Antin JH, Ritz J, Dubovsky JA, Byrd JC, MacDonald KP, Hill GR, Blazar BR. Increased T follicular helper cells and germinal center B cells are required for cGVHD and bronchiolitis obliterans. Blood. 2014 Jun 19;123(25):3988-98. doi: 10.1182/blood-2014-03-562231. Epub 2014 May 12. PMID 24820310
- [Result] Weiss JM, Chen W, Nyuydzefe MS, Trzeciak A, Flynn R, Tonra JR, Marusic S, Blazar BR, Waksal SD, Zanin-Zhorov A. ROCK2 signaling is required to induce a subset of T follicular helper cells through opposing effects on STATs in autoimmune settings. Sci Signal. 2016 Jul 19;9(437):ra73. doi: 10.1126/scisignal.aad8953. PMID 27436361